CLINICAL TRIAL: NCT02368340
Title: A Longitudinal Study of Hermansky-Pudlak Syndrome Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: University of South Florida (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lisa Young, Associate Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 150104; U54HL127672 (NIH)
Record Dates: First submitted 2015-02-13; First posted 2015-02-23 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Hermansky Pudlak Syndrome
MeSH Terms: conditions — Hermanski-Pudlak Syndrome | interventions — Respiratory Physiological Phenomena; Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, lymphocytes
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Adults with pulmonary fibrosis: This group includes adults with HPS who have known pulmonary fibrosis. Subjects in this group will provide blood and urine specimens.
  Interventions: Other: Sample collection
- Adults at-risk: This group includes adults with HPS with subtypes at-risk for pulmonary fibrosis, but who do not have known pulmonary fibrosis.
  Subjects in this group will undergo chest CT and pulmonary function testing, and provide blood and urine specimens.
  Interventions: Other: Pulmonary function test; Other: Chest CT; Other: Sample collection
- HPS adults not at-risk: This group includes adults with HPS subtypes considered not at-risk for pulmonary fibrosis.
  Subjects in this group will provide blood and urine specimens.
  Interventions: Other: Sample collection
- Children with HPS at-risk: This group includes children with HPS subtypes at-risk for pulmonary fibrosis. Subjects in this group will undergo pulmonary function testing, and provide blood and urine specimens.
  Interventions: Other: Pulmonary function test; Other: Sample collection

INTERVENTIONS:
Other: Pulmonary function test — Pulmonary function testing performed
  Groups: Adults at-risk; Children with HPS at-risk
Other: Chest CT — Chest CT scan to evaluate for pulmonary fibrosis
  Groups: Adults at-risk
Other: Sample collection — Blood and urine sample collections

SUMMARY:
Hermansky-Pudlak Syndrome (HPS) is a rare genetic disease that is associated with oculocutaneous albinism, bleeding, granulomatous colitis, and pulmonary fibrosis in some subtypes, including HPS-1, HPS-2, and HPS-4. Pulmonary fibrosis causes shortness of breath and progressive decline in lung function. In HPS patients with at-risk subtypes, almost all adults eventually develop fatal pulmonary fibrosis unless they undergo lung transplantation.

The purpose of this study is to identify the earliest measurable pulmonary disease activity in individuals at-risk for HPS pulmonary fibrosis. The study also aims to develop biomarkers that will aid in understanding of the causes of HPS pulmonary fibrosis and facilitate more rapid conduct of therapeutic trials in HPS patients with mild pulmonary disease in the future.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ages 12-90 years with confirmed diagnosis of HPS as defined by verification of reduced or absent platelet dense granules by electron microscopy and/or genetic diagnosis
* Ability to provide informed consent, or consent of parent/guardian and assent for minors

Exclusion Criteria:

* Status-post lung transplantation
* Perceived unsuitability for participation in the study in the opinion of the investigator

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with diagnosis of Hermansky-Pudlak Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Chest CT scan | change in CT Scan from baseline to 2.5 years

SECONDARY OUTCOMES:
Pulmonary function test | change in PFTs from baseline to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R. Young, MD, Principal Investigator — Vanderbilt University
Locations (5):
- United States (5):
  - Loyola University Medical Center, Maywood, Illinois
  - Brigham and Women's Hospital, Harvard, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee